CLINICAL TRIAL: NCT04099355
Title: Investigating the Effect of Dronabinol on Post-surgical Pain
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Psychiatrist II, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7815
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Knee Replacement; Arthropathy of Knee
MeSH Terms: interventions — Dronabinol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dronabinol (Experimental): active group
  Interventions: Drug: Dronabinol 5mg Cap; Drug: Non-active comparator
- control (Placebo Comparator): control group
  Interventions: Drug: Dronabinol 5mg Cap; Drug: Non-active comparator

INTERVENTIONS:
Drug: Dronabinol 5mg Cap — 1 QAM and 2 QHS PO 14 days
Drug: Non-active comparator — 1 QAM and 2 QHS PO 14 days

SUMMARY:
This study is designed to investigate the effect of dronabinol on post operative pain in patients undergoing total knee replacement (for their own clinical care).

DETAILED DESCRIPTION:
Total knee replacement is a common surgical procedure that restores function to the damaged joint. Recovery from this procedure takes weeks and requires opioids to manage post-surgical pain. The goal of this study is to investigate whether dronabinol (synthetic THC) can reduce pain and the need for opioid medication following this particular surgery.

Subjects will be recruited from the Department of Orthopedic Surgery. All subjects will undergo total knee replacement as part of their clinical care (the surgery itself is not part of this study). The study begins following discharge from the hospital. They will be asked to take dronabinol or placebo as they recover from surgery. During this time they will be given their usual pain medications at discharge which includes opioids for pain. The opioids are to be taken if the subject is experiencing pain. The investigator's hypothesis is that subjects taking dronabinol will need fewer doses of opioids to control pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing total knee arthroplasty (TKA) at the CUIMC department of orthopedic surgery as part of their clinical care.
* Able to give informed consent and comply with study procedures in English

Exclusion Criteria:

* Meet DSM-V criteria for current major psychiatric illness, such as bipolar disorder, major depression, or psychosis. Subjects with a current substance use disorder will be excluded. Subjects with a past cannabis use disorder are excluded.
* Diagnosis of a major medical or neurological disorder, including orthostatic hypertension, cardiovascular disease (congestive heart failure, unstable angina, or a history of cardiac infarction), hypotension, or neurodegenerative disorders.
* Subjects taking medications that can lead to a drug interaction.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form | 2 weeks
  pain assessment, self report measure of pain, scale 0-10 (10 worst)

SECONDARY OUTCOMES:
opioid medication log | two weeks
  opioid use by participant for pain after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, MD, Principal Investigator — NYSPI
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No